CLINICAL TRIAL: NCT04136444
Title: An Open-Label, Parallel-Group, Pharmacokinetic Study of Padsevonil in Study Participants With Either Normal Hepatic Function or With Moderately Impaired Hepatic Function (Child-Pugh Class B)
Brief Title: A Pharmacokinetic Study of Padsevonil in Study Participants With Either Normal or Moderately Impaired Hepatic Function
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Based on available data, UCB has decided to stop development of padsevonil as adjunctive treatment of focal-onset seizures
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UP0056
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Results first posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Healthy Study Participants; Impaired Hepatic Function
Keywords: Padsevonil; Phase 1; Pharmacokinetic; PSL
MeSH Terms: interventions — padsevonil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy participants (Experimental): Participants will receive assigned single and multiple doses of padsevonil.
  Interventions: Drug: Padsevonil
- Hepatically impaired participants (Experimental): Participants will receive assigned single and multiple doses of padsevonil.
  Interventions: Drug: Padsevonil

INTERVENTIONS:
Drug: Padsevonil — Padsevonil will be administered in predefined dosages.
  Other Names: PSL; UCB0942

SUMMARY:
The purpose of the study is to evaluate the plasma pharmacokinetic (PK), safety and tolerability of padsevonil (PSL) in hepatically impaired and non-hepatically impaired study participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be male or female 18 to 70 years of age, inclusive, at the time of signing the informed consent
* Participant must have body weight of at least 50 kg (males) or 45 kg (females) and body mass index within the range 18 to 38 kg/m^2 (inclusive)
* Participants must meet the following requirements to be included in the study:

  1. A male participant must agree to use contraception during both Treatment Periods and for at least 7 days after the last dose of study medication and refrain from donating sperm during this period
  2. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies:

     Not a woman of childbearing potential (WOCBP) OR A WOCBP who agrees to follow the contraceptive guidance during both Treatment Periods and for at least 90 days (or 5 terminal half-lives) after the final dose of study medication

     Specific inclusion criteria for study participants WITH moderate hepatic insufficiency:
* Participant must have characteristics that will meet the clinical criteria usually found in participants with chronic hepatic insufficiency, as determined by medical history and physical examinations (eg, echography, scintigraphy, biopsy, or some specific laboratory values as evidence)

Exclusion Criteria:

* Participant has any medical or psychiatric condition that, in the opinion of the Investigator, could jeopardize or compromise the study participant's ability to participate in this study, such as a history of schizophrenia, or other psychotic disorder, bipolar disorder, or severe unipolar depression. The presence of potential psychiatric exclusion criteria will be determined based on the psychiatric history collected at Screening Visit
* Participant has a known hypersensitivity to any components of the study medication as stated in this protocol
* Participant has a lifetime history of suicide attempt (including an actual attempt, interrupted attempt, or aborted attempt), or has had suicidal ideation in the past 6 months
* Participant has past or intended use of over-the-counter or prescription medication including herbal remedies and hepatic enzyme inhibitors within 2 weeks or 5 half-lives prior to dosing, particularly for participants with hepatic impairment where t1/2 may be prolonged. Specific medications may be allowed. Participant has used hepatic enzyme-inducing drugs (eg, glucocorticoids, phenobarbital, phenytoin, isoniazid, or rifampicin, etc.) within 2 months prior to dosing unless required to treat an adverse event (AE). This does not include oral contraceptives not exceeding 30 μg ethinyl estradiol or postmenopausal hormone replacement therapy (HRT) or implants, patches, or intrauterine devices (IUDs) /intrauterine systems (IUSs) delivering progesterone (for female study participants) or acetaminophen with a maximal dose of 2 g/day or with a maximum of 10g over 15 days. In case of uncertainty, the UCB Study Physician should be consulted
* Participant has a history of chronic alcohol or drug abuse within the previous 12 months. Participant has a positive pre-study drug/alcohol screen (to include at minimum: amphetamines, barbiturates, cocaine, opiates, cannabinoids, and benzodiazepines). A participant with a positive finding on the drug screen may still be enrolled at the discretion of the Investigator if a plausible clinical explanation exists (eg, prior or concomitant medication use)
* Participant has a history of unexplained syncope or a family history of sudden death due to long QT syndrome
* Participant has renal impairment as indicated by an estimated glomerular filtration rate (GFR) <60 mL/min, calculated by using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI)
* Participant tests positive for human immunodeficiency virus-1/2 antibody (HIV-1/2Ab) at Screening or within 3 months prior to the first dose of study medication

Specific exclusion criteria for study participants WITHOUT hepatic insufficiency

* Participant has alanine aminotransferase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase (ALP) >1.0x upper limit of normal (ULN)
* Participant has bilirubin >1.0xULN (isolated bilirubin >1.0xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Participant has current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones) Note: For participants with a Baseline result >ULN for ALT, AST, ALP, or total bilirubin, a baseline diagnosis and/or the cause of any clinically meaningful elevation must be understood and recorded in the electronic Case Report Form (eCRF). If participant has >ULN ALT, AST, or ALP that does not meet the exclusion limit at Screening, repeat the tests, if possible, prior to dosing to ensure there is no further ongoing clinically relevant increase. In case of a clinically relevant increase, inclusion of the study participant must be discussed with the UCB Study Physician

Specific exclusion criteria for study participants WITH moderate hepatic insufficiency

* Participant has acute liver failure of any etiology
* Participant has biliary cirrhosis
* Participant has used any drug indicated for the medical care of moderate hepatic insufficiency that is not established in dose and schedule for at least 14 days before the first liver function test (except paracetamol with a maximal dose of 2 g/day or with a maximum of 10 g over 15 days)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (1):
- Up0056 004, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, Individual Patient Data cannot be adequately anonymized and there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll study participants in October 2019 and concluded in May 2020.
Pre-assignment Details: Participant Flow refers to the Safety Set (SS).
Groups:
- Cohort A: Healthy study participants in Cohort A received a single dose of padsevonil 100 milligrams (mg) on Day 1 of Treatment Period 1 and multiple doses of padsevonil 100 mg twice daily (bid) from Day 8 to 11 and a single dose of padsevonil 100 mg on Day 12 during Treatment Period 2 as oral tablets. There was a Washout Period of 6 days between Treatment Period 1 and 2.
- Cohort B: Participants with moderate hepatic insufficiency in Cohort B received a single dose of padsevonil 100 mg on Day 1 of Treatment Period 1 and multiple doses of padsevonil 100 mg bid from Day 8 to 11 and a single dose of padsevonil 100 mg on Day 12 during Treatment Period 2 as oral tablets. There was a Washout Period of 6 days between Treatment Period 1 and 2.
Period: Overall Study
Arm/Group | Cohort A | Cohort B
Started | 3 | 9
Completed | 3 (The cohort was not completely recruited, as the study was stopped/terminated due to COVID-19.) | 8
Not Completed | 0 | 1
Not completed — Sponsor request due to undisclosed concomitant medication | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set (SS) which consisted of all study participants who received at least 1 dose of the investigational medicinal product (IMP).
Arm/Group | Cohort A | Cohort B | Total Title
Number analyzed (Participants) | 3 | 9 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 9 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (7.5) | 57.8 (4.3) | 57.6 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 1 | 6 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 2 | 2
  White | 3 | 7 | 10

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of a Single Dose Padsevonil (PSL)
Description: Cmax is maximum observed plasma concentration.
Time Frame: Plasma samples were taken predose on Day 1 and 0.25, 0.5, 0.75, 1, 1.5, 3, 4, 5, 6, 8, 12, 24, 48, 72 and 96 hours postdose
Population: The Pharmacokinetic Set (PKS) is a subset of the Full Analysis Set (FAS), consisting of those study participants who had no important protocol deviations affecting the PK parameters and had a sufficient number of samples available to determine at least 1 PK parameter. All PK analyses were performed using the PKS.
Measure: Geometric Mean (95% Confidence Interval); unit: nanograms/milliliter (ng/mL)
Groups:
- Cohort A (PKS): Healthy study participants in Cohort A received a single dose of padsevonil 100 mg on Day 1 of Treatment Period 1 and multiple doses of padsevonil 100 mg bid from Day 8 to 11 and a single dose of padsevonil 100 mg on Day 12 during Treatment Period 2 as oral tablets. Participants formed the Pharmacokinetic Set (PKS).
- Cohort B (PKS): Participants with moderate hepatic insufficiency in Cohort B received a single dose of padsevonil 100 mg on Day 1 of Treatment Period 1 and multiple doses of padsevonil 100 mg bid from Day 8 to 11 and a single dose of padsevonil 100 mg on Day 12 during Treatment Period 2 as oral tablets. There was a Washout Period of 6 days between Treatment Period. Participants formed the PKS.
Arm/Group | Cohort A (PKS) | Cohort B (PKS)
Number analyzed (Participants) | 3 | 8
nanograms/milliliter (ng/mL) | NA [NA to NA] — As pre-specified in the Protocol/Statistical Analysis Plan, Geometric Means are only calculated if at least 2/3 of the individual data points are above lower limit of quantification (LLOQ). | 531.4 [347.5 to 812.7]

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to t (AUC0-t) of a Single Dose Padsevonil (PSL)
Description: AUC (0-t) is defined as area under the plasma concentration-time curve from time zero to time t.
Time Frame: as for outcome 1
Population: The Pharmacokinetic Set (PKS) is a subset of the FAS, consisting of those study participants who had no important protocol deviations affecting the PK parameters and had a sufficient number of samples available to determine at least 1 PK parameter. All PK analyses were performed using the PKS.
Measure: Geometric Mean (95% Confidence Interval); unit: hours*nanograms per milliliter (h*ng/mL)
Arm/Group | Cohort A (PKS) | Cohort B (PKS)
Number analyzed (Participants) | 3 | 8
hours*nanograms per milliliter (h*ng/mL) | NA [NA to NA] — As pre-specified in the Protocol/Statistical Analysis Plan, Geometric Means are only calculated if at least 2/3 of the individual data points are above LLOQ. | 3793 [1896 to 7591]

3. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC) From Time 0 to Infinity of a Single Dose Padsevonil (PSL)
Description: AUC is defined as area under the plasma concentration-time curve from time 0 to infinity.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: hours*ng/mL
Arm/Group | Cohort A (PKS) | Cohort B (PKS)
Number analyzed (Participants) | 3 | 8
hours*ng/mL | NA [NA to NA] — As pre-specified in the Protocol/Statistical Analysis Plan, Geometric Means are only calculated if at least 2/3 of the individual data points are above LLOQ. | 3830 [1911 to 7677]

4. Primary Outcome: Maximum Observed Plasma Concentration at Steady-state (Cmax,ss) of Multiple Doses Padsevonil (PSL)
Description: Cmax,ss is defined as maximum observed plasma concentration at steady-state.
Time Frame: On Days 8, 9, 10 and 11 PK samples were taken predose. On Day 12, PK samples were taken predose and 0.25, 0.5, 0.75, 1, 1.5, 3, 4, 5, 6, 8, 12, 24 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: nanograms per milliliter (ng/mL)
Arm/Group | Cohort A (PKS) | Cohort B (PKS)
Number analyzed (Participants) | 3 | 8
nanograms per milliliter (ng/mL) | NA [NA to NA] — As pre-specified in the Protocol/Statistical Analysis Plan, Geometric Means are only calculated if at least 2/3 of the individual data points are above LLOQ. | 558.1 [346.9 to 897.8]

5. Primary Outcome: Area Under the Concentration-time Curve (AUCtau) at Steady-state Over a Dosing Interval of Multiple Doses Padsevonil (PSL)
Description: AUCtau is defined as area under the curve over a dosing interval at steady-state.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: hours*ng/mL
Arm/Group | Cohort A (PKS) | Cohort B (PKS)
Number analyzed (Participants) | 3 | 8
hours*ng/mL | NA [NA to NA] — As pre-specified in the Protocol/Statistical Analysis Plan, Geometric Means are only calculated if at least 2/3 of the individual data points are above LLOQ. | 3783 [2260 to 6332]

6. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. A treatment-emergent adverse event was characterized according to the intake of the study medication.
Time Frame: From Baseline until End of Study Visit (up to Day 18)
Population: The Safety Set (SS) consisted of all study participants who received at least 1 dose of the investigational medicinal product (IMP). Study participants were classified according to the treatment that was actually received. All safety analyses were performed using the SS.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A Single Dose (SS): Healthy study participants in Cohort A received a single dose of padsevonil 100 mg on Day 1 of Treatment Period 1 as oral tablets. Participants formed the Safety Set (SS).
- Cohort B Single Dose (SS): Participants with moderate hepatic insufficiency in Cohort B received a single dose of padsevonil 100 mg on Day 1 of Treatment Period 1 as oral tablets. Participants formed the SS.
- Cohort A Multiple Dose (SS): Healthy study participants in Cohort A received multiple doses of padsevonil 100 mg bid from Day 8 to 11 and a single dose of padsevonil 100 mg on Day 12 during Treatment Period 2 as oral tablets. Participants formed the SS.
- Cohort B Multiple Dose (SS): Participants with moderate hepatic insufficiency in Cohort B received multiple doses of padsevonil 100 mg bid from Day 8 to 11 and a single dose of padsevonil 100 mg on Day 12 during Treatment Period 2 as oral tablets. Participants formed the SS.
Arm/Group | Cohort A Single Dose (SS) | Cohort B Single Dose (SS) | Cohort A Multiple Dose (SS) | Cohort B Multiple Dose (SS)
Number analyzed (Participants) | 3 | 9 | 3 | 9
Participants | 3 | 6 | 3 | 7

7. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: A serious adverse event (SAE) is any untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Requires in patient hospitalization or prolongation of existing hospitalization
  * Is a congenital anomaly or birth defect
  * Is an infection that requires treatment parenteral antibiotics
  * Other important medical events which based on medical or scientific judgement may jeopardize the patients, or may require medical or surgical intervention to prevent any of the above.
Time Frame: From Baseline until End of Study Visit (up to Day 18)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A Single Dose (SS) | Cohort B Single Dose (SS) | Cohort A Multiple Dose (SS) | Cohort B Multiple Dose (SS)
Number analyzed (Participants) | 3 | 9 | 3 | 9
Participants | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Leading to Discontinuation of the Study
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. A treatment-emergent adverse event was characterized according to the intake of the study medication. TEAEs leading to discontinuation of the study are reported.
Time Frame: From Baseline until End of Study Visit (up to Day 18)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A Single Dose (SS) | Cohort B Single Dose (SS) | Cohort A Multiple Dose (SS) | Cohort B Multiple Dose (SS)
Number analyzed (Participants) | 3 | 9 | 3 | 9
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent Adverse Events (AEs) were collected from Baseline until End of Study Visit (up to Day 18)
Description: Treatment-emergent AE was defined as any AE with a start date/time on or after the first dose of study medication or any unresolved event already present before administration of study medication that worsened in intensity following exposure to the treatment.
Arm/Group | Cohort A Single Dose (SS) | Cohort B Single Dose (SS) | Cohort A Multiple Dose (SS) | Cohort B Multiple Dose (SS)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/9 | 0/3 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/9 | 0/3 | 0/9
Other Adverse Events (participants affected / at risk) | 3/3 | 6/9 | 3/3 | 7/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A Single Dose (SS) (N=3) | Cohort B Single Dose (SS) (N=9) | Cohort A Multiple Dose (SS) (N=3) | Cohort B Multiple Dose (SS) (N=9)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Clumsiness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 3 (3) | 2 (2) | 3 (3) | 3 (3)
Bradyphrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-07-02): https://cdn.clinicaltrials.gov/large-docs/44/NCT04136444/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-26): https://cdn.clinicaltrials.gov/large-docs/44/NCT04136444/SAP_001.pdf